CLINICAL TRIAL: NCT00207558
Title: Blood Folate and Homocysteine Levels Following Administration of Folic Acid According to Different Daily Dosing Schedules:a Simulation of Food Fortification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Peking University (Other); Ministry of Science and Technology of the People´s Republic of China (Other Government); University of Florida (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CDC-NCBDDD-3970; U11/CCU015587-04-1; U11/CCU015586-05
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2006-07-13 (Estimated); Status verified 2005-09

CONDITIONS: Neural Tube Defects - Spina Bifida and Anencephaly
MeSH Terms: conditions — Anencephaly | interventions — Folic Acid

INTERVENTIONS:
Drug: folic acid

SUMMARY:
The aim of this study is to examine whether the same total daily dosage of folic acid, when taken as a single daily dose or as multiple divided doses throughout the day, results in different blood folate and homocysteine levels at the conclusion of the study. Further, a comparison of blood folate and homocysteine levels among women taking daily low-dosage (100mcg) and standard- dosage (400mcg) folic acid with those of women taking daily or weekly high-dosage (4000mcg) folic acid will be conducted.

ELIGIBILITY:
Inclusion Criteria:

-women who have delivered a baby two to four years ago, whose child is still alive, who are not breast-feeding, who are not pregnant or planning to become pregnant within the next 9 months following enrollment, who are using an IUD for contraception, and who have not taken vitamin supplements during the past 3 months

Exclusion Criteria:

-women who have not delivered a baby two to four years ago, whose child is deceased, who are breast-feeding, who are currently pregnant or planning to become pregnant within the next 9 months following enrollment, who are not using an IUD for contraception, and who have taken vitamin supplements during the past 3 months

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1100

CONTACTS AND LOCATIONS:
Locations (1):
- Townships, Xianghe County, Hebei, China

REFERENCES:
- [Derived] Chen MY, Rose CE, Qi YP, Williams JL, Yeung LF, Berry RJ, Hao L, Cannon MJ, Crider KS. Defining the plasma folate concentration associated with the red blood cell folate concentration threshold for optimal neural tube defects prevention: a population-based, randomized trial of folic acid supplementation. Am J Clin Nutr. 2019 May 1;109(5):1452-1461. doi: 10.1093/ajcn/nqz027. PMID 31005964
- [Derived] Crider KS, Zhu JH, Hao L, Yang QH, Yang TP, Gindler J, Maneval DR, Quinlivan EP, Li Z, Bailey LB, Berry RJ. MTHFR 677C->T genotype is associated with folate and homocysteine concentrations in a large, population-based, double-blind trial of folic acid supplementation. Am J Clin Nutr. 2011 Jun;93(6):1365-72. doi: 10.3945/ajcn.110.004671. Epub 2011 Apr 20. PMID 21508090